CLINICAL TRIAL: NCT02968004
Title: A Phase 3, Open-label, Randomized, Multicenter, 12 Months, Efficacy and Safety Study of Weekly MOD-4023 Compared to Daily Genotropin - Therapy in Pre-pubertal Children With Growth Hormone Deficiency
Brief Title: Safety and Efficacy Phase 3 Study of Long-acting hGH (MOD-4023) in Growth Hormone Deficient Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-4-006
Record Dates: First submitted 2016-11-13; First posted 2016-11-18 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Growth Hormone Deficiency
MeSH Terms: interventions — MOD-4023; somatrogon; Human Growth Hormone

ARMS (2):
- MOD-4023 (Experimental): Once weekly subcutaneous injection of long acting r-hGH (MOD-4023)
  Interventions: Drug: MOD-4023
- Genotropin (Active Comparator): Once daily subcutaneous injection of somatropin (r-hGH; Genotropin)
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: MOD-4023 — Once weekly subcutaneous injection using pre-filled pen device.
  Other Names: Somatrogon
  Arms: MOD-4023
Drug: Somatropin — Once daily subcutaneous injection of Genotropin using pre-filled pen device.
  Other Names: Genotropin
  Arms: Genotropin

SUMMARY:
This is an open-label, randomized, multicenter, efficacy and safety study of weekly MOD-4023 compared to daily Genotropin therapy in pre-pubertal children with growth hormone deficiency.

DETAILED DESCRIPTION:
The study consists of a 12 month, open-label, randomized, active controlled, parallel group study comparing the efficacy and safety of weekly MOD-4023 to daily growth hormone (GH), Genotropin. After 12 months, subjects will have the option to enter the long term open-label extension.

ELIGIBILITY:
Main Study Inclusion Criteria:

1. Pre-pubertal children aged ≥3 years, and not yet 11 years for girls or not yet 12 years for boys with either isolated GHD, or GH insufficiency as part of multiple pituitary hormone deficiency.
2. Confirmed diagnosis of GHD by two different GH provocation tests defined as a peak plasma GH level of ≤10 ng/mL.
3. Bone age (BA) is not older than chronological age and should be less than 10 for girls and less than 11 for boys.
4. Without prior exposure to any r-hGH therapy (naïve patients).
5. Impaired height and height velocity defined as:

   * Annualized height velocity (HV) below the 25th percentile for CA (HV < -0.7 SDS) and gender according to sponsor calculator
   * The interval between 2 height measurements should be at least 6 months, but should not exceed 18 months prior to inclusion
6. Baseline IGF-1 level of at least 1 SD below the mean IGF-1 level standardized for age and sex (IGF-1 SDS ≤-1)
7. Normal calculated GFR per updated bedside Schwartz formula for pediatric patients.
8. Children with multiple hormonal deficiencies must be on stable replacement therapies (no change in dose) for other hypothalamo-pituitary-organ axes for at least 3 months prior ICF signing.
9. Normal 46XX karyotype for girls.
10. Willing and able to provide written informed consent of the parent or legal guardian and written assent from patient.

    LT-OLE Inclusion Criteria:
11. Completion of the main study (12 months of treatment) with adequate compliance.
12. Willing and able to provide written informed consent of the parent or legal guardian and written assent from patient.
13. Agree to refrain from sexual activity.

Main Study Exclusion Criteria:

1. Children with prior history of leukemia, lymphoma, sarcoma or any other forms of cancer.
2. History of radiation therapy or chemotherapy.
3. Malnourished children defined as BMI < -2 SDS for age and sex.
4. Children with psychosocial dwarfism.
5. Children born small for gestational age (SGA - birth weight and/or birth length <-2 SDS for gestational age).
6. Presence of anti-hGH antibodies at screening.
7. Any clinically significant abnormality likely to affect growth or the ability to evaluate growth, such as, but not limited to, chronic diseases like renal insufficiency, spinal cord irradiation, etc.
8. T2 and T1 diabetic patients, who in the opinion of the investigator are not receiving standard of care treatment or are non-compliant with their prescribed treatment or who are in poor metabolic control.
9. Chromosomal abnormalities including Turner's syndrome, Laron syndrome, Noonan syndrome, Prader-Willi syndrome, Russell-Silver syndrome, SHOX mutations/deletions and skeletal dysplasias.
10. Concomitant administration of other treatments that may have an effect on growth such as anabolic steroids, or sex steroids, with the exception of ADHD drugs or hormone replacement therapies (thyroxin, hydrocortisone, desmopressin).
11. Children requiring glucocorticoid therapy (e.g. for asthma) that are taking chronically a dose greater than 400 μg/d of inhaled budesonide or equivalent.
12. Major medical conditions and/or presence of contraindication to r-hGH treatment.
13. More than one closed epiphyses.
14. Known or suspected HIV-positive patient, or patient with advanced diseases such as AIDS or tuberculosis.
15. Drug, substance, or alcohol abuse.
16. Known hypersensitivity to the components of study medication.
17. Other causes of short stature such as celiac disease, uncontrolled primary hypothyroidism and rickets.
18. Likely non-compliance in respect to study conduct.
19. Participation in any other trial of an investigational agent within 30 days prior to consent.
20. Study enrollment has been met or study is closed by sponsor prior to completion of screening process.

    LT-OLE Exclusion Criteria:
21. Concomitant administration of other treatments that may have an effect on growth such as anabolic steroids, or sex steroids, with the exception of ADHD drugs or HRT (thyroxin, hydrocortisone, desmopressin).
22. Change in medical condition during the treatment period (such as, but not limited to, development of a serious inter-current critical illness, a severe adverse drug reaction, etc.).
23. Positive pregnancy test.
24. Unresolved drug related (Genotropin or MOD-4023) SAE from the treatment period as per medical monitor judgement.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2016-12; Primary Completion 2019-08 (Actual); Study Completion 2024-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Cruz, Study Director — Sponsor GmbH
Locations (81):
- United States (18):
  - Children's Hospital of Orange County- Children's Clinic, Orange, California
  - Children's Hospital- Colorado, Aurora, Colorado
  - Rocky Mountain Pediatrics, Centennial, Colorado
  - Nemours Children's Health System, Jacksonville, Florida
  - University of Miami Medical Center, Miami, Florida
  - St Luke's Children's Specialty Center, Boise, Idaho
  - Children's Hospital of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - University of Massachusettes, Worcester, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - The Diabetes & Obesity Clinical Specialist, Las Vegas, Nevada
  - Goryeb Children's Hospital, Morristown, New Jersey
  - Buffalo Children's Hospital, Buffalo, New York
  - Albert Einstein College of Medicine at Yeshiva University, Mineola, New York
  - Children's Hospital of Cincinnati / Cincinnati Center for Growth Disorders, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
  - Mary Bridge Children's Hospital & Health Center, Tacoma, Washington
- Argentina (2):
  - Hospital Materno Infantil San Roque, Paraná, Entre Ríos Province
  - Hospital de Ninos de la Santisima Trinidad Cordoba, Córdoba
- Australia (3):
  - John Hunter Children's Hospital, New Lambton Heights, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - PM Hospital for Children, Subiaco, Western Australia
- Health Institution- 2nd City Pediatric Hospital, Minsk, Belarus
- MHAT Sveta Marina, Varna, Bulgaria
- Centre de recherche du CHU Sainte-Justine, Montreal, Quebec, Canada
- Colombia (3):
  - Dexa Diab, Bogotá
  - Uniendo, Bogotá
  - Hospital Pablo Tobon Uribe, Medellín
- Georgia (2):
  - Maritime Hospital JSC, Batumi
  - Vere XXI JSC, Tbilisi
- Greece (2):
  - Aghia Sophia Children's Hospital, Athens
  - General Children's Hospital of Athens P&A Kyriakou, Athens
- India (8):
  - Manipal Hospital, Bengaluru, Karnataka
  - Getwell Health & Research Institute, Nagpur, Maharashtra
  - Jehangir Clinical Development Centre, Pune, Maharashtra
  - Postgraduate Institute of Medical Education and Research, Chandigarh, Punjab
  - Care Hospital, Hyderabad, Telangna
  - Meditrina Institute of Medical Sciences, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Sir Gangaram Hospital, New Delhi
- Israel (9):
  - Haemek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Assaf Harofeh Medical Center, Be’er Ya‘aqov
  - Bnei Zion Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Scheider Children's Medical Center, Petah Tikva
  - Tel Hashomer Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv
- Hospital Angeles de Puebla, Puebla City, Reserva Territorial Atilxcayotl, Mexico
- New Zealand (2):
  - The Liggins Institute, Grafton, Auckland
  - Wellington Children's Hospital, Newtown, Wellington Region
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne in Gdansk, Gdansk
  - Centrum Zdrowia Matki Polki, Lodz
- Russia (6):
  - Bashkirian State Medical University, Ufa, Bashlortostan Republic
  - Kazan State Medical Univeristy/Pediatric Republic Clinical Hospital, Kazan', Tatarstan Republic
  - Endocrinology Scientific Center, Moscow
  - Pediatric City Clinical Hospital/Russian Medical Academy of Continuous Education, Moscow
  - Saint Petersburg State Pediatric Medical University, Saint Petersburg
  - Voronezh State Medical University, Voronezh
- South Korea (5):
  - Bundang Cha Hospital, Seongnam-si, Gyeonggi-do
  - Inje University Busan Paik Hospital, Busan
  - KyungPook National University Hospital, Daegu
  - Chosun University Hospital, Gwangju
  - Severance Hospital, Seoul
- Spain (6):
  - Hospital Miguel Servet, Zaragoza, Aragon
  - Hospital Josep Trueta, Girona, Catalonia
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo
  - Parc Tauli, Sabadell
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Ukraine (5):
  - Ukrainian Research and Practical Centre of Endocrine Surgery, Transplantation of Endocrine Organs and Tissues of the Ministry of Health of Ukraine, Kyiv
  - Institute of Endocrinology and Metabolism/VP Komisarenko of Academy of Medical Science of Ukraine, Kyiv
  - Odesa Regional Clinical Children's Hospital, Odesa
  - Vinnitsa Regional Clinical Highly Specialized Endocrinology Centre, Vinnitsa
  - Zaporizhzhya Regional Clinical Child Hospital, Zaporizhzhya
- United Kingdom (2):
  - Royal Hospital for Children, Glasgow
  - St. George's University Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomez R, Khadilkar V, Shembalkar J, Chu DM, Ko CW, Wajnrajch MP, Wang R. Post hoc subgroup analysis of Asian children with paediatric GHD from the global phase 3 efficacy and safety study of once-weekly somatrogon vs. once-daily somatropin. J Pediatr Endocrinol Metab. 2024 May 9;37(6):525-531. doi: 10.1515/jpem-2023-0512. Print 2024 Jun 25. PMID 38717038
- [Derived] Loftus J, Quitmann J, Valluri SR. Health-related quality of life in pre-pubertal children with pediatric growth hormone deficiency: 12-month results from a phase 3 clinical trial of once-weekly somatrogon versus once-daily somatropin. Curr Med Res Opin. 2024 Feb;40(2):175-184. doi: 10.1080/03007995.2023.2290623. Epub 2024 Jan 24. PMID 38053515
- [Derived] Gomez R, Lamoureux R, Turner-Bowker DM, Loftus J, Maghnie M, Miller BS, Polak M, Yaworsky A. Physician experience with once-weekly somatrogon versus once-daily rhGH regimen in pediatric patients with growth hormone deficiency: a cross-sectional survey of physicians from the global phase 3 study. Front Endocrinol (Lausanne). 2023 Oct 17;14:1254424. doi: 10.3389/fendo.2023.1254424. eCollection 2023. PMID 37955005
- [Derived] Deal CL, Steelman J, Vlachopapadopoulou E, Stawerska R, Silverman LA, Phillip M, Kim HS, Ko C, Malievskiy O, Cara JF, Roland CL, Taylor CT, Valluri SR, Wajnrajch MP, Pastrak A, Miller BS. Efficacy and Safety of Weekly Somatrogon vs Daily Somatropin in Children With Growth Hormone Deficiency: A Phase 3 Study. J Clin Endocrinol Metab. 2022 Jun 16;107(7):e2717-e2728. doi: 10.1210/clinem/dgac220. PMID 35405011

RESULTS

PARTICIPANT FLOW:
Groups:
- MOD-4023: Once weekly subcutaneous injection of long acting r-hGH (MOD-4023)
  MOD-4023: Once weekly subcutaneous injection using pre-filled pen device.
  Note that in the OLE Phase of the study all subjects were treated with MOD-4023. The distribution noted across different arms is in reference to the assigned drug during the Main Study Phase.
- Genotropin: Once daily subcutaneous injection of somatropin (r-hGH; Genotropin)
  Somatropin: Once daily subcutaneous injection of Genotropin
  Note that in the OLE Phase of the study all subjects were treated with MOD-4023. The distribution noted across different arms is in reference to the assigned drug during the Main Study Phase.
Period: Main Study Phase
Arm/Group | MOD-4023 | Genotropin
Started | 109 | 115
Completed | 108 | 114
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Open Label Extension (OLE) Year 1
Arm/Group | MOD-4023 | Genotropin
Started | 104 (Of 109 participants entered the Main Study Phase, 4 completed the study and 1 discontinued. Therefore, 104 entered the OLE period Year 1.) | 108 (Of 115 participants entered the Main Study Phase, 6 completed the study and 1 discontinued. Therefore, 108 entered the OLE period Year 1.)
Completed | 102 | 99
Not Completed | 2 | 9
Not completed — Adverse Event | 0 | 6
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Miscellaneous | 0 | 1
Period: Open Label Extension (OLE) Year 2
Arm/Group | MOD-4023 | Genotropin
Started | 91 (Of 104 participants entered the OLE period Year 1, 11 completed the study and 2 discontinued. Therefore, 91 entered the OLE period Year 2.) | 86 (Of 108 participants entered the OLE period Year 1, 13 completed the study and 9 discontinued. Therefore, 86 entered the OLE period Year 2.)
Completed | 88 | 82
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Miscellaneous | 0 | 1
Period: Open Label Extension (OLE) Year 3
Arm/Group | MOD-4023 | Genotropin
Started | 88 (Of 91 participants entered the OLE period Year 2, 3 discontinued. Therefore, 88 entered the OLE period Year 3.) | 82 (Of 86 participants entered the OLE period Year 2, 4 discontinued. Therefore, 82 entered the OLE period Year 3.)
Completed | 84 | 80
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Prohibited Treatments | 0 | 1
Not completed — Local Crisis | 1 | 0
Period: Open Label Extension (OLE) Year 4
Arm/Group | MOD-4023 | Genotropin
Started | 83 (Of 88 participants entered the OLE period Year 3, 1 completed the study and 4 discontinued. Therefore, 83 entered the OLE period Year 4.) | 79 (Of 82 participants entered the OLE period Year 3, 1 completed the study and 2 discontinued. Therefore, 79 entered the OLE period Year 4.)
Completed | 38 | 43
Not Completed | 45 | 36
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Non-Compliance With Study Drug | 0 | 1
Not completed — Sponsor Discontinuation of Study | 27 | 21
Not completed — Bone Age Reached | 3 | 1
Not completed — Local Crisis | 10 | 9
Not completed — Miscellaneous | 2 | 0
Period: Open Label Extension (OLE) Year 5
Arm/Group | MOD-4023 | Genotropin
Started | 24 (Of 83 participants entered the OLE period Year 4, 14 completed the study and 45 discontinued. Therefore, 24 entered the OLE period Year 5.) | 28 (Of 79 participants entered the OLE period Year 4, 15 completed the study and 36 discontinued. Therefore, 28 entered the OLE period Year 5.)
Completed | 18 | 22
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Sponsor Discontinuation of Study | 2 | 6
Not completed — Bone Age Reached, | 1 | 0
Not completed — Closure of Epiphyseal Plates | 1 | 0
Not completed — Local Crisis | 1 | 0
Period: Open Label Extension (OLE) Year 6
Arm/Group | MOD-4023 | Genotropin
Started | 0 (Of 24 participants entered the OLE period Year 5, 18 completed the study and 6 discontinued. Therefore, 0 entered the OLE period Year 6.) | 2 (Of 28 participants entered the OLE period Year 5, 20 completed the study and 6 discontinued. Therefore, 2 entered the OLE period Year 6.)
Completed | 0 | 0
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Genotropin: Once daily subcutaneous injection of somatropin (r-hGH; Genotropin)
  Somatropin: Once daily subcutaneous injection of Genotropin
- Total: Total of all reporting groups
Arm/Group | MOD-4023 | Genotropin | Total
Number analyzed (Participants) | 109 | 115 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.83 (2.66) | 7.61 (2.37) | 7.72 (2.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 36 | 63
  Male | 82 | 79 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 24
  Not Hispanic or Latino | 98 | 102 | 200
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 81 | 86 | 167
  Black or African American | 0 | 2 | 2
  Asian | 24 | 21 | 45
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 3 | 5 | 8
  Unknown | 0 | 0 | 0
  Multiracial | 0 | 0 | 0
  Not reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Colombia | 4 | 4 | 8
  Argentina | 1 | 2 | 3
  United States | 17 | 25 | 42
  Ukraine | 13 | 11 | 24
  United Kingdom | 0 | 3 | 3
  Belarus | 1 | 1 | 2
  India | 12 | 14 | 26
  Russia | 8 | 12 | 20
  Spain | 10 | 9 | 19
  Greece | 3 | 0 | 3
  New Zealand | 3 | 1 | 4
  Canada | 3 | 2 | 5
  South Korea | 8 | 4 | 12
  Turkey | 1 | 0 | 1
  Taiwan | 0 | 2 | 2
  Poland | 7 | 12 | 19
  Mexico | 2 | 0 | 2
  Georgia | 5 | 1 | 6
  Israel | 7 | 8 | 15
  Australia | 2 | 2 | 4
  Bulgaria | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Annual Height Velocity in Main Study Phase
Description: Annual Height Velocity in cm. Annual Height Velocity at 12 months is based on the difference between the heights at 12 months and baseline.
Time Frame: 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/year
Arm/Group | MOD-4023 | Genotropin
Number analyzed (Participants) | 109 | 115
cm/year | 10.10 [9.58 to 10.63] | 9.78 [9.29 to 10.26]

2. Primary Outcome: Annual Height Velocity in OLE Phase
Description: Annualized Height Velocity (cm/year) in OLE Phase
Time Frame: Up to 60 months
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | MOD-4023 | Genotropin
Number analyzed (Participants) | 104 | 108
cm/year
  OLE Month 0 | 10.27 (2.38) | 9.72 (2.50)
  OLE Month 12: number analyzed (Participants) | 91 | 82
  OLE Month 12 | 8.03 (1.81) | 8.21 (1.87)
  OLE Month 24: number analyzed (Participants) | 89 | 84
  OLE Month 24 | 7.78 (1.91) | 8.05 (1.77)
  OLE Month 36: number analyzed (Participants) | 83 | 79
  OLE Month 36 | 6.90 (1.80) | 7.14 (1.69)
  OLE Month 48: number analyzed (Participants) | 34 | 41
  OLE Month 48 | 6.19 (1.62) | 6.86 (2.08)
  OLE Month 60: number analyzed (Participants) | 0 | 4
  OLE Month 60 |  | 5.05 (1.10)

3. Secondary Outcome: Height Velocity at 6 Months in Main Study Phase
Description: Height velocity in cm measured after 6 months of treatment. Annualized Height velocity after 6 months is calculated based on the difference between the heights at 6 months and baseline.
Time Frame: After 6 months of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/year
Arm/Group | MOD-4023 | Genotropin
Number analyzed (Participants) | 109 | 115
cm/year | 10.59 [9.96 to 11.22] | 10.04 [9.47 to 10.62]

4. Secondary Outcome: Change in Height Standard Deviation Score (SDS) in Main Study Phase
Description: Change in height Standard Deviation Score (SDS) after 6 and 12 months is calculated based on the difference between the heights at 6 and 12 months and baseline.
Time Frame: After 6 and 12 months
Population: Two subjects discontinued, one from each group.
Measure: Mean (95% Confidence Interval); unit: Standard Deviation Score
Arm/Group | MOD-4023 | Genotropin
Number analyzed (Participants) | 109 | 115
Standard Deviation Score
  SDS at 6 months | 0.54 [0.48 to 0.61] | 0.48 [0.42 to 0.54]
  SDS at 12 months | 0.92 [0.82 to 1.02] | 0.87 [0.78 to 0.96]

5. Secondary Outcome: Change in Bone Maturation (BM) in Main Study Phase
Description: Annual change in bone age measurements as per Gruelich-Pyle method
Time Frame: 52 weeks
Population: 5 participants of MOD-4023 and 13 participants of Genotropin did not have bone age measurements at 12 months.
Measure: Mean (Standard Deviation); unit: ratio of bone age to chronologic age
Arm/Group | MOD-4023 | Genotropin
Number analyzed (Participants) | 104 | 102
ratio of bone age to chronologic age | 0.05 (0.09) | 0.06 (0.1)

6. Secondary Outcome: Insulin-like Growth Factor-1 (IGF-1) Standard Deviation Score (SDS) in Main Study Phase
Description: Via central lab analysis
Time Frame: Baseline and at 12 months
Population: 2 subjects in MOD-4023 and 5 subjects in Genotropin didn't have the measurements at 12 months
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS)
Arm/Group | MOD-4023 | Genotropin
Number analyzed (Participants) | 109 | 115
Standard Deviation Score (SDS)
  Baseline | -1.95 (0.89) | -1.72 (0.90)
  At 12 months: number analyzed (Participants) | 107 | 110
  At 12 months | 0.65 (1.32) | -0.69 (1.09)

7. Secondary Outcome: Change in Height Standard Deviation Score (SDS) in OLE Phase
Description: Change in height Standard Deviation Score (SDS) at each time point is calculated based on the difference between the time point and baseline.
Time Frame: 60 months
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Standard Deviation Score
Arm/Group | MOD-4023 | Genotropin
Number analyzed (Participants) | 104 | 108
Standard Deviation Score
  Baseline (from Main Study Phase) | -2.95 (1.30) | -2.79 (1.31)
  OLE Month 0 | 0.95 (0.55) | 0.85 (0.52)
  OLE Month 12: number analyzed (Participants) | 91 | 82
  OLE Month 12 | 1.38 (0.78) | 1.34 (0.71)
  OLE Month 24: number analyzed (Participants) | 89 | 84
  OLE Month 24 | 1.57 (0.77) | 1.66 (0.78)
  OLE Month 36: number analyzed (Participants) | 83 | 79
  OLE Month 36 | 1.81 (0.85) | 1.93 (0.85)
  OLE Month 48: number analyzed (Participants) | 34 | 41
  OLE Month 48 | 1.96 (0.67) | 2.04 (0.81)
  OLE Month 60: number analyzed (Participants) | 0 | 4
  OLE Month 60 |  | 2.14 (0.38)

8. Secondary Outcome: Insulin-like Growth Factor-1 (IGF-1) Standard Deviation Score (SDS) in OLE Phase
Time Frame: 60 Months
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Standard Deviation Score
Arm/Group | MOD-4023 | Genotropin
Number analyzed (Participants) | 104 | 108
Standard Deviation Score
  Baseline (from Main Study Phase) | 77.91 (46.11) | 83.10 (41.17)
  OLE Month 0: number analyzed (Participants) | 97 | 105
  OLE Month 0 | 185.9 (107.1) | 69.96 (59.92)
  OLE Month 12: number analyzed (Participants) | 83 | 86
  OLE Month 12 | 255.9 (120.0) | 248.6 (111.9)
  OLE Month 24: number analyzed (Participants) | 76 | 80
  OLE Month 24 | 293.4 (132.8) | 295.3 (137.5)
  OLE Month 36: number analyzed (Participants) | 73 | 76
  OLE Month 36 | 315.6 (139.7) | 330.7 (138.0)
  OLE Month 48: number analyzed (Participants) | 29 | 38
  OLE Month 48 | 354.8 (133.1) | 368.9 (124.9)
  OLE Month 60: number analyzed (Participants) | 0 | 4
  OLE Month 60 |  | 397.5 (85.27)

9. Other Pre Specified Outcome: Device
Description: Proportion of successful single injections out of total number of single injections using the MOD-4023 Pen in the USA
Time Frame: 6 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Device
Description: Proportion of successful single injections out of total number of single injections using the MOD-4023 Pen in the USA at Week 1 based on the Observer Assessment Tool (OAT)
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | MOD-4023
Number analyzed (Participants) | 17
Participants | 17

ADVERSE EVENTS:
Time Frame: 1 year for Main Study Phase. Up to 6 years for OLE Phase.
Groups:
- MOD-4023 in OLE Phase: Once weekly subcutaneous injection of long acting r-hGH (MOD-4023)
  MOD-4023: Once weekly subcutaneous injection using pre-filled pen device.
Arm/Group | MOD-4023 | Genotropin | MOD-4023 in OLE Phase
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/115 | 0/212
Serious Adverse Events (participants affected / at risk) | 3/109 | 2/115 | 14/212
Other Adverse Events (participants affected / at risk) | 92/109 | 90/115 | 175/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MOD-4023 (N=109) | Genotropin (N=115) | MOD-4023 in OLE Phase (N=212)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 1
Delayed Puberty (Endocrine disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Noninfective Sialoadenitis (Gastrointestinal disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 4
Croup Infectious (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 1
Chronic tonsillitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Scrotal Varicose Veins (Reproductive system and breast disorders) | 0 | 0 | 1
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Kawasaki's Disease (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MOD-4023 (N=109) | Genotropin (N=115) | MOD-4023 in OLE Phase (N=212)
Anaemia (Blood and lymphatic system disorders) | 7 | 7 | 5
Basophilia (Blood and lymphatic system disorders) | 0 | 0 | 6
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 11
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 1
Ear Pain (Ear and labyrinth disorders) | 2 | 7 | 7
Hypothyroidism (Endocrine disorders) | 7 | 3 | 12
Conjunctivitis Allergic (Eye disorders) | 3 | 0 | 2
Myopia (Eye disorders) | 0 | 0 | 6
Abdominal Pain (Gastrointestinal disorders) | 4 | 2 | 9
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 6 | 12
Constipation (Gastrointestinal disorders) | 2 | 4 | 5
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 14
Nausea (Gastrointestinal disorders) | 3 | 1 | 6
Toothache (Gastrointestinal disorders) | 0 | 0 | 6
Vomiting (Gastrointestinal disorders) | 8 | 9 | 23
Injection Site Erythema (General disorders) | 9 | 0 | 11
Injection Site Induration (General disorders) | 4 | 1 | 2
Injection Site Pain (General disorders) | 43 | 29 | 66
Injection Site Pruritus (General disorders) | 6 | 0 | 6
Injection Site Swelling (General disorders) | 5 | 0 | 6
Pyrexia (General disorders) | 18 | 16 | 40
Vaccination Site Pain (General disorders) | 0 | 0 | 5
Seasonal Allergy (Immune system disorders) | 0 | 0 | 6
Bronchitis (Infections and infestations) | 3 | 9 | 15
Conjunctivitis (Infections and infestations) | 3 | 3 | 4
Corona Virus Infection (Infections and infestations) | 0 | 0 | 37
Enterobiasis (Infections and infestations) | 4 | 2 | 4
Gastroenteritis (Infections and infestations) | 4 | 3 | 8
Gastroenteritis Viral (Infections and infestations) | 0 | 3 | 4
Influenza (Infections and infestations) | 5 | 3 | 22
Molluscum Contagiosum (Infections and infestations) | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 25 | 29 | 66
Otitis Externa (Infections and infestations) | 4 | 4 | 3
Otitis Media (Infections and infestations) | 4 | 7 | 9
Otitis Media Acute (Infections and infestations) | 1 | 3 | 3
Pharyngitis (Infections and infestations) | 7 | 5 | 7
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 7
Pneumonia (Infections and infestations) | 0 | 0 | 5
Rhinitis (Infections and infestations) | 6 | 1 | 10
Sinusitis (Infections and infestations) | 0 | 0 | 5
Tonsillitis (Infections and infestations) | 5 | 6 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 7
Viral Infection (Infections and infestations) | 0 | 0 | 5
Viral Pharyngitis (Infections and infestations) | 0 | 0 | 5
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 12
Arthropod Bite (Injury, poisoning and procedural complications) | 6 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 5
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 7
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 6
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 6
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 5
Blood Creatine Phosphokinase Increased (Investigations) | 2 | 8 | 3
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 | 3 | 1
Coronavirus Test Positive (Investigations) | 0 | 0 | 15
Free Fatty Acids Increased (Investigations) | 5 | 1 | 11
Insulin-Like Growth Factor Increased (Investigations) | 0 | 0 | 5
Low Density Lipoprotein Decreased (Investigations) | 0 | 0 | 5
Thyroxine Free Decreased (Investigations) | 0 | 0 | 7
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Hypoinsulinaemia (Metabolism and nutrition disorders) | 4 | 3 | 6
Iron Deficiency (Metabolism and nutrition disorders) | 1 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 8 | 10
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 10
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 8
Headache (Nervous system disorders) | 18 | 25 | 41
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 0 | 0 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 24
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 8
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 18
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 12
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 4
Rash generalised (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT02968004/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT02968004/SAP_002.pdf